CLINICAL TRIAL: NCT02872532
Title: Testicular Tissue Cryopreservation for Fertility Preservation in Males Facing Fertility Threatening Diagnoses or Treatment Regimens
Brief Title: Testicular Tissue Cryopreservation in Children
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Candace F. Granberg, M.D., Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15-004891; NCI-2022-10961 (Registry Identifier: CTRP (Clinical Trials Reporting Program))
Record Dates: First submitted 2016-08-16; First posted 2016-08-19 (Estimated); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Cancer; Cancer-Related Condition; Infertility
MeSH Terms: conditions — Neoplasms; Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Testicular tissue (Experimental): Children faced with a fertility threatening diagnosis or treatment plan will be offered testicular tissue cryopreservation, particularly if pre-pubescent and without other options to preserve fertility.
  Interventions: Procedure: Testicular tissue cryopreservation

INTERVENTIONS:
Procedure: Testicular tissue cryopreservation — Testicular tissue will be removed

SUMMARY:
This protocol is being designed to offer testicular tissue cryopreservation to male pediatric patients (0-17 years of age) with fertility threatening medical diagnoses or facing surgery, chemotherapy or radiation therapy that may cause loss of reproductive potential.

DETAILED DESCRIPTION:
Testicular tissue cryopreservation is currently considered experimental but offers the only opportunity for fertility preservation in pre-pubescent boys faced with a fertility threatening diagnosis or treatment plan.

After completion of study intervention, patients are followed up at 1-week post-surgery and then yearly thereafter.

ELIGIBILITY:
Inclusion Criteria: (All inclusion criteria must be met.)

* Be male 0-17 years of age
* Meet at least one of the following four conditions:

  * Be scheduled to undergo surgery, chemotherapy, drug treatment and/or radiation for the treatment or prevention of a medical condition or malignancy with risk of causing permanent and complete loss of subsequent testicular function. Risk categories based on treatment regimens are indicated below. Investigators will utilize three sources to calculate risk: 1. "Fertile Hope - Risks of Azoospermia" brochure that details typical agents and treatment regimens in each risk category, 2. The Summed Alkylating Agent dose score (Green et al., 2009) or 3. The Cyclophosphamide Equivalent Dose method (Green et al., 2014). Because of the complexity of many treatment regimens, patient risk categorization will be at the discretion of the investigators.

    * High Risk

      * >= 80% risk of prolonged azoospermia, Fertile Hope Brochure
      * Summed alkylating agent dose score >= 3
      * Cyclophosphamide equivalent dose >= 7,500mg/m^2
    * Intermediate risk (21-79% risk of prolonged azoospermia, Fertile Hope)
    * Low Risk ( =< 20% risk of prolonged azoospermia, Fertile Hope)
    * Eligibility is limited to patients in the High risk category and/or intermediate risk after discussion with pediatric oncology, fertility preservation team, and the patient/family
  * Or, have a medical condition or malignancy that requires removal of all or part of one or both testicles
  * Or, have a medical condition (genetic or autoimmune) that results in decline in fertility (e.g. Klinefelter syndrome)
  * Or, have a newly diagnosed or recurrent disease affecting fertility. Those who were not enrolled at the time of initial diagnosis (i.e. patients with recurrent disease) are eligible if they have not previous received therapy that is viewed as likely to result in complete and permanent loss of testicular function
* Have two testicles if undergoing elective removal of a testicle for fertility preservation only. Note: removal of both testicles will limit fertility preservation options. Or have 1 testicle but limited potential for future fertility due to underlying condition, malignancy, prior surgery or previous torsion and no other fertility preservation methods are available except for testicular tissue cryopreservation
* Sign an approved informed consent and authorization permitting the release of personal health information. The patient and/or the patient's legally authorized guardian must acknowledge in writing that consent for specimen collection has been obtained, in accordance with institutional policies approved by the United States (U.S.) Department of Health and Human Services
* Consent for serum screening tests for infectious diseases to be performed at the time of testicular tissue harvesting. The immediate testing will include but not be limited to testing for Hepatitis B, Hepatitis C, and human immunodeficiency virus (HIV)
* Undergo a full history and physical examination and obtain standard pre-operative clearance (based on the most recent American College of Cardiology/ American Heart Association [ACC/AHA] Guideline for Perioperative Cardiovascular Evaluation for Noncardiac Surgery) as determined by their primary surgeon
* Note: In cases of torsion of testicles or other medical conditions that result in impairment of testicular function, patients can be consented and included in the study, if during the testicular surgery the provider finds that the patient still has viable tissue that can be cryopreserved.

Exclusion Criteria: (Any exclusion criteria will disqualify.)

* Diagnosed with psychological, psychiatric, or other conditions which prevent giving fully informed consent.
* Diagnosed with an underlying medical condition that significantly increases their risk of complications from anesthesia and surgery.
* Previous recipients of gonadotoxic chemotherapy or radiation therapy thought to have resulted in impairment of testicular function.

Ages: 0 Years to 17 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2016-08-16 (Actual); Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Number of pregnancies and live births after transplantation of cryopreserved testicular tissue | 10-20 years

CONTACTS AND LOCATIONS:
Overall Officials: Candace F. Granberg, MD, Principal Investigator — Mayo Clinic in Rochester
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Joshi VB, Behl S, Pittock ST, Arndt CAS, Zhao Y, Khan Z, Granberg CF, Chattha A. Establishment of a Pediatric Ovarian and Testicular Cryopreservation Program for Malignant and Non-Malignant Conditions: The Mayo Clinic Experience. J Pediatr Adolesc Gynecol. 2021 Oct;34(5):673-680. doi: 10.1016/j.jpag.2021.04.006. Epub 2021 Apr 25. PMID 33910089
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials